CLINICAL TRIAL: NCT00212888
Title: A Pilot Study to Determine the Impact of Therapeutic HIV Vaccination Followed by a Scheduled Interruption of Antiretroviral Therapy on HIV-Specific Immune Function and Virologic Rebound in Patients With Prolonged Viral Suppression
Brief Title: Combination Vaccination Before HIV Treatment Interruption
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario HIV Treatment Network (Network); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000456-01H; CTA file 9427-C1574-32C
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: HIV Infections
Keywords: HIV; Vaccination
MeSH Terms: conditions — HIV Infections | interventions — remune; ALVAC vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Remune and ALVAC — * Group 1) Remune™ (1ml i.m.) at weeks 0, 12 and 20 and ALVAC (1 ml i.m.) at weeks 8, 12, 16 and 20);
  * Group 2) Remune™ placebo (1ml i.m.) at weeks 0, 12 and 20 and ALVAC (1 ml i.m.) at weeks 8, 12, 16 and 20; or
  * Group 3) Remune™ placebo (1ml i.m.) at weeks 0, 12 and 20 and ALVAC placebo (1 ml i.m.) at weeks 8, 12, 16 and 20.

SUMMARY:
The purpose of this study is to determine if vaccination before a structured treatment interruption (STI) is associated with an improvement in immune function, resulting in a delayed and reduced rebound in the amount of HIV virus in the blood.

DETAILED DESCRIPTION:
Volunteers will be randomly assigned to receive the vaccines or matching placebos before interrupting their antiretroviral therapy at week 24.

Dosage:

Remune(TM) 1 ml i.m.* at weeks 0, 12, and 20; ALVAC 1 ml i.m.* at weeks 8,12, 16, and 20.

* i.m.: injected in a muscle

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection (by serology)
* HIV RNA level below 50 copies/ml for at least two years
* Receiving at least 2 antiretroviral agents including at least 1 protease inhibitor or 1 non-nucleoside reverse transcriptase inhibitor at time of screening
* Have CD4 counts above 500 cells/ul
* Have CD4/CD8 ratio above 0.5
* Have never had a CD4 count below 250
* No previous AIDS-defining opportunistic infection
* No previous cancer chemotherapy or other system immunosuppressive therapy (excluding brief courses [<= 1 month] of prednisone or its equivalent)
* Able to provide informed consent

Exclusion Criteria:

* Hepatitis B surface antigen positive
* Hepatitis C antibody positive
* AST, ALT, ALP, creatinine, urea above three times the normal upper limit
* Blood abnormalities (hemoglobin lower than 100, white blood cell count [WBC] lower than 1500 or platelets lower than 100)
* Allergies to components of Remune™ or ALVAC
* Contraindications to vaccine components
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-04; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Angel, MD, Principal Investigator — OHRI
Locations (3):
- Canada (3):
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - CHUM Hotel-Dieu, Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec

REFERENCES:
- [Derived] Angel JB, Routy JP, Tremblay C, Ayers D, Woods R, Singer J, Bernard N, Kovacs C, Smaill F, Gurunathan S, Sekaly RP. A randomized controlled trial of HIV therapeutic vaccination using ALVAC with or without Remune. AIDS. 2011 Mar 27;25(6):731-9. doi: 10.1097/QAD.0b013e328344cea5. PMID 21330911

RESULTS

PARTICIPANT FLOW:
Groups:
- ALVAC With Remune: Remune™ (1ml i.m.) at weeks 0, 12 and 20 and ALVAC (1 ml i.m.) at weeks 8, 12, 16 and 20.
- ALVAC With Remune Placebo: Remune™ placebo (1ml i.m.) at weeks 0, 12 and 20 and ALVAC (1 ml i.m.) at weeks 8, 12, 16 and 20.
- Both Placebos: Remune™ placebo (1ml i.m.) at weeks 0, 12 and 20 and ALVAC placebo (1 ml i.m.) at weeks 8, 12, 16 and 20.
Period: Overall Study
Arm/Group | ALVAC With Remune | ALVAC With Remune Placebo | Both Placebos
Started | 19 | 18 | 15
Completed | 16 | 18 | 14
Not Completed | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALVAC With Remune | ALVAC With Remune Placebo | Both Placebos | Total
Number analyzed (Participants) | 19 | 18 | 15 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39.7 [32.2 to 45.8] | 41.5 [35.7 to 49.6] | 43.4 [39.3 to 48.2] | 41.8 [37.3 to 47.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 12
  Male | 15 | 13 | 12 | 40
Duration on ART [Median (Inter-Quartile Range); unit: years] | 3.61 [2.47 to 5.92] | 5.15 [2.98 to 7.08] | 5.18 [3.51 to 8.11] | 4.89 [2.85 to 6.87]
Baseline CD4 cell count [Median (Inter-Quartile Range); unit: cells/ul] | 771 [660 to 970] | 658 [514 to 1029] | 848 [576 to 953] | 768 [568 to 957]
Baseline CD4% [Median (Inter-Quartile Range); unit: percent] | 37.1 [34.0 to 45.0] | 38.0 [32.0 to 42.2] | 35.0 [31.9 to 43.5] | 37.2 [32.2 to 43.2]
CD4 nadir [Median (Inter-Quartile Range); unit: cells/ul] | 347 [259 to 454] | 326 [272 to 482] | 368 [277 to 497] | 353 [268 to 462]
Pre-HAART HIV-RNA [Median (Inter-Quartile Range); unit: log 10 (copies/ml)] | 4.4 [3.5 to 5.0] | 4.0 [3.1 to 4.4] | 4.2 [3.6 to 5.2] | 4.1 [3.6 to 4.8]
Presence of 'protective' HLA allele [Number; unit: participants] — Protective HLA alleles include B27, B57, B58
  participants | 3 | 2 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time to Detectable Virus in the Remune Plus ALVAC Group and the Placebo Group
Time Frame: Up to week 48
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ALVAC With Remune | Both Placebos
Number analyzed (Participants) | 16 | 14
days | 24.5 [11 to 32] | 13.5 [11 to 25]

2. Secondary Outcome: Time to Detectable Virus in the ALVAC Alone Group and the Placebo Group
Time Frame: Up to week 48
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ALVAC With Remune Placebo | Both Placebos
Number analyzed (Participants) | 18 | 14
days | 23.0 [16 to 31] | 13.5 [11 to 25]

3. Secondary Outcome: Time to Rebound of Plasma HIV RNA Level to 10,000 Copies/ml
Time Frame: Up to week 48
Population: Only participants who reached 10,000 copies/ml are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ALVAC With Remune | ALVAC With Remune Placebo | Both Placebos
Number analyzed (Participants) | 13 | 15 | 12
days | 30.0 [18 to 44] | 31.0 [25 to 37] | 24.5 [21 to 30]

4. Secondary Outcome: Viral Set-point
Description: Viral set-point is the viral load (HIV RNA) that the body settles at within a few weeks to months after infection with HIV.
Time Frame: Up to week 48
Population: Only participants whose viral loads reached a steady state are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: log10 copies/ml
Arm/Group | ALVAC With Remune | ALVAC With Remune Placebo | Both Placebos
Number analyzed (Participants) | 14 | 17 | 12
log10 copies/ml | 4.4 [3.4 to 4.7] | 4.2 [3.8 to 4.4] | 4.5 [3.8 to 5.2]

5. Secondary Outcome: Magnitude of Viral Rebound
Description: Magnitude of viral rebound is the amount of HIV viral load an infected person who was previously on ART and suppressed below clinical detection rebounds to following ART stoppage. This will typically be compared to the viral load before starting ART or Viral set-point discussed earlier.
Time Frame: Up to week 48
Measure: Median (Inter-Quartile Range); unit: log10 copies/ml
Arm/Group | ALVAC With Remune | ALVAC With Remune Placebo | Both Placebos
Number analyzed (Participants) | 16 | 18 | 14
log10 copies/ml | 4.8 [4.2 to 5.2] | 5.0 [4.3 to 5.4] | 5.0 [4.6 to 5.6]

6. Secondary Outcome: HIV-specific Immune Function
Time Frame: at week 48
Population: Data not collected for this assessment.
Arm/Group | ALVAC With Remune | ALVAC With Remune Placebo | Both Placebos
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | ALVAC With Remune | ALVAC With Remune Placebo | Both Placebos
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 12/19 | 10/18 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALVAC With Remune (N=19) | ALVAC With Remune Placebo (N=18) | Both Placebos (N=15)
Injection site reaction (Skin and subcutaneous tissue disorders) | 7 | 9 | 3
Subjective fever (General disorders) | 5 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes